CLINICAL TRIAL: NCT07338578
Title: Comparison of Propofol and Sevoflurane in Terms of Hemodynamics and Bronchoscopist Satisfaction in Patients Who Underwent Endobronchial Ultrasound Guided Transbronchial Needle Aspiration Under General Anesthesia
Brief Title: A Study Comparing Sevoflurane and Propofol in Patients Undergoing Endobronchial Ultrasound Guided Needle Aspiration
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: SBU-HAMIDIYE-23-57
Record Dates: First submitted 2025-11-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Hemodynamic Stability; Pulmonary Diseases or Conditions; Complication of Anesthesia
Keywords: EBUS; Propofol; Sevoflurane; Outpatient Anesthesia; General Anesthesia
MeSH Terms: conditions — Lung Diseases | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Propofol Group: Group 1: Patients who received total intravenous anesthesia (TIVA) with propofol during EBUS-TBNA.
  Interventions: Drug: propofol
- Group 2: Sevoflurane Group: Patients who received inhalational anesthesia with sevoflurane during EBUS-TBNA.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: propofol — In group 1, anesthesia was induced intravenously and maintained using propofol to achieve an adequate depth of anesthesia and hemodynamic stability during EBUS- TBNA. The airway was managed with a size 4 laryngeal mask airway (LMA) allowing bronchoscope insertion and controlled ventilation. Standard monitoring included ECG, noninvasive blood pressure, pulse oximetry, and capnography.
  Other Names: Diprivan
  Groups: Group 1: Propofol Group
Drug: Sevoflurane — In group 2, following intravenous induction, anesthesia was maintained using sevoflurane in an oxygen-air mixture to ensure adequate depth of anesthesia and hemodynamic stability during EBUS-TBNA. Airway management was achieved using a size 4 laryngeal mask airway (LMA) to facilitate bronchoscope insertion and controlled ventilation. Standard monitoring included ECG, noninvasive blood pressure, pulse oximetry, and capnography.
  Other Names: Sevorane
  Groups: Group 2: Sevoflurane Group

SUMMARY:
Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is a minimally invasive procedure used to obtain samples from mediastinal and hilar lymph nodes or lung parenchymal lesions for diagnostic and staging purposes. The success and safety of the procedure, including diagnostic yield, complication rates, and bronchoscopist comfort, depend largely on the choice of anesthesia technique. General anesthesia is frequently preferred because it provides a stable airway, adequate ventilation, and improved procedural conditions.

Patient-related factors such as medical status, history, procedure duration, and number of needle passes may influence hemodynamic stability and tolerance, making anesthesiologist involvement essential. Previous studies comparing intravenous and inhalational anesthesia in various surgical and bronchoscopic procedures have evaluated their effects on hemodynamics, complications, recovery time, visibility of the surgical field, and postoperative outcomes. However, there is limited evidence directly comparing propofol-based total intravenous anesthesia and sevoflurane-based inhalational anesthesia specifically for EBUS-TBNA.

This study aims to compare the effects of propofol and sevoflurane anesthesia on perioperative hemodynamic parameters, respiratory stability, and procedure-related complications in patients undergoing EBUS-TBNA. In addition, the study assesses bronchoscopist satisfaction with each anesthetic technique, including procedural comfort and working conditions. The findings are expected to contribute to optimizing anesthetic management for EBUS-TBNA, improving patient safety, and enhancing procedural quality.

DETAILED DESCRIPTION:
This prospective, single-center, observational cohort study was designed to compare the effects of two general anesthesia techniques-propofol based total intravenous anesthesia (TIVA) and sevoflurane based inhalational anesthesia-on hemodynamic parameters and bronchoscopist satisfaction in patients undergoing endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA).

EBUS-TBNA is a minimally invasive bronchoscopic procedure that allows tissue sampling from mediastinal and hilar lymph nodes or pulmonary nodules. The procedure plays a major role in the diagnosis and staging of lung cancer and other mediastinal pathologies. Although EBUS-TBNA has become an established diagnostic tool with a high safety profile, anesthetic management during the procedure remains a matter of debate. Appropriate anesthesia choice affects not only patient safety and comfort but also the bronchoscopist's technical performance.

Patients scheduled for EBUS-TBNA under general anesthesia were included after obtaining institutional ethics approval. Individuals aged 18 years or older with American Society of Anesthesiologists (ASA) physical status I-III were eligible. Exclusion criteria included incomplete medical records, combined surgical interventions, severe hemodynamic instability, or ASA class IV or higher. All patients provided written informed consent prior to the procedure.

The study population was divided into two groups according to the anesthetic technique used. In the Sevoflurane Group, anesthesia was induced with intravenous agents and maintained using inhalational sevoflurane in a mixture of oxygen and air. In the Propofol Group, anesthesia was maintained with continuous intravenous infusion of propofol. In both groups, anesthesia depth was monitored clinically and adjusted to maintain stable hemodynamics and adequate oxygenation. All procedures were performed with the patient in the supine position under controlled ventilation using a size 4 laryngeal mask airway (LMA), chosen for its ability to maintain a secure airway and allow sufficient space for bronchoscopic manipulation.

Standard monitoring included continuous electrocardiography, noninvasive blood pressure measurement, pulse oximetry, and capnography. Hemodynamic parameters such as heart rate, mean arterial pressure (MAP), oxygen saturation (SpO₂), and end-tidal CO₂ (EtCO₂) were recorded at baseline (pre-induction), after induction, during bronchoscope insertion, at 5-minute intervals during the procedure, and immediately after completion. The total doses of anesthetic and vasoactive drugs, as well as the need for supplemental medications, were documented.

At the end of the procedure the occurrence of complications such as hypoxia, bronchospasm, coughing, or airway trauma were also noted. The bronchoscopist, blinded to the anesthetic regimen, evaluated procedural satisfaction immediately after each case using a standardized satisfaction scale (graded as poor, fair, good, or excellent). Factors considered included surgical field stability, visibility, and patient movement.

The primary outcome measure of the study was hemodynamic stability, assessed through changes in mean arterial pressure and heart rate between groups. Secondary outcome measures included bronchoscopist satisfaction, airway related complications. Descriptive statistics were used for demographic and procedural variables. Intergroup comparisons were performed using Student's t-test or Mann-Whitney U test for continuous variables and chi-square or Fisher's exact test for categorical variables. A p-value < 0.05 was considered statistically significant.

The results of this study are expected to provide evidence regarding the relative advantages and limitations of propofol and sevoflurane anesthesia in EBUS-TBNA procedures. Understanding how each anesthetic technique affects intraoperative stability and procedural comfort can help optimize anesthetic management strategies, improve patient safety, and enhance bronchoscopist performance in minimally invasive airway interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years) with an ASA physical status I-III who provided written informed consent were included.

Exclusion Criteria:

* ASA ≥ IV
* chronic cough or dyspnea
* preoperative desaturation (SpO₂ < 90%)
* hypotension (MAP < 60 mmHg),
* bradycardia (HR < 60 bpm),
* hypersensitivity to anesthetics,
* any form of organ failure,
* laboratory abnormalities (electrolyte imbalance, anemia, polycythemia, thrombocytosis, leukopenia, or leukocytosis),
* perioperative hypo- or hyperthermia, dehydration, or overhydration.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients who underwent endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) under general anesthesia at a tertiary training and research hospital. All participants were scheduled for diagnostic bronchoscopy for evaluation of pulmonary or mediastinal lesions. Patients with American Society of Anesthesiologists (ASA) physical status I-III were included.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure During EBUS-TBNA | Periprocedural period (from anesthesia induction to 60 minutes after procedure completion)
  Systolic blood pressure (mmHg) will be measured at baseline (pre-induction), immediately after induction, during the procedure at 5-minute intervals, at the end of the procedure, and upon arrival in the recovery room. Values will be compared between the propofol and sevoflurane groups.
Change in Diastolic Blood Pressure During EBUS-TBNA | Periprocedural period (from anesthesia induction to 60 minutes after procedure completion)
  Diastolic blood pressure (mmHg) will be measured at baseline (pre-induction), immediately after induction, during the procedure at 5-minute intervals, at the end of the procedure, and upon arrival in the recovery room. Values will be compared between the propofol and sevoflurane groups.
Change in Heart Rate During EBUS-TBNA | Periprocedural period (from anesthesia induction to 60 minutes after procedure completion)
  Heart rate (beats per minute) will be recorded at baseline (pre-induction), immediately after induction, during the procedure at 5-minute intervals, at the end of the procedure, and upon arrival in the recovery room. Values will be compared between the propofol and sevoflurane groups.
Bronchoscopist Satisfaction Score During EBUS-TBNA | Immediately after completion of the procedure.
  Bronchoscopist satisfaction will be assessed using a standardized 5-point Likert scale, where higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
Procedure-Related Complications | During the procedure and up to 1 hour postoperatively.
  To record and compare the incidence of complications such as hypoxia, bronchospasm, cough, laryngospasm, airway trauma, and postoperative nausea or vomiting between the two anesthesia techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Sari, MD, Principal Investigator — University of Health Sciences, Sultan 2. Abdulhamid Han Training and Research Hospital; Tuna Erturk, MD, Study Chair — University of Health Sciences, Sultan 2. Abdulhamid Han Training and Research Hospital; Suheyla Abitagaoglu, MD, Study Chair — University of Health Sciences, Sultan 2. Abdulhamid Han Training and Research Hospital
Locations (1):
- University of Health Sciences, Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data include patient-specific clinical information collected under institutional ethics approval and are intended for internal research analysis only. Summary results may be shared in scientific publications and presentations.